CLINICAL TRIAL: NCT00005482
Title: Homocyst(e)Ine, Vitamin Status, and CVD Risk
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4969; R01HL054711 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Cerebrovascular Accident; Coronary Disease; Myocardial Infarction; Heart Diseases; Hyperhomocysteinemia
MeSH Terms: conditions — Cardiovascular Diseases; Stroke; Coronary Disease; Myocardial Infarction; Heart Diseases; Hyperhomocysteinemia

SUMMARY:
To test the hypotheses that the risk of myocardial infarction and/or stroke is associated with elevated plasma levels of homocysteine, and low plasma levels of folate, vitamins B12 and B6.

DETAILED DESCRIPTION:
BACKGROUND:

Elevated plasma homocyst(e)ine is a risk factor for vascular disease in middle-aged men. Supplementation with folate, and to some extent vitamins B12 and B6, can reduce plasma homocyst(e)ine levels. There is also evidence from in vitro studies that the adverse atherogenic or thrombotic effects of Lp(a) may be greatly enhanced by homocyst(e)ine. The high prevalence of low levels of folate and vitamins B12 and B6 among the elderly in the United States has led to the hypothesis that a substantial portion of cardiovascular morbidity and mortality among older persons could be prevented by increasing intake of these nutrients to reduce plasma levels of homocysteine. Little is known, however, regarding the relationship of homocysteine, folate, B vitamins, and Lp(a) to cardiovascular disease among the elderly, among whom CVD represents the leading cause of morbidity and mortality.

DESIGN NARRATIVE:

In this ancillary study to the prospective Cardiovascular Health Study (CHS), a case-cohort design was used to test hypotheses that the risk of myocardial infarction and/or stoke was associated with elevated plasma levels of homocysteine, and low plasma levels of folate, vitamins B12 and B6. Further, a determination was made whether elevated plasma levels of homocysteine and Lp(a) interacted to increase substantially the risk of myocardial infarction and/or stroke above that due to either factor alone. The sub-cohort was used to study the relationship between the factors under study and progression of sub-clinical atherosclerosis. For each case and sub-cohort member, an aliquot of fasting plasma drawn at baseline was analyzed for homocysteine, folate B12, and B6 concentrations. [Values of plasma Lp(a) were determined at baseline.] Results of these assays were combined with other CHS data to address the hypothesis that the risk of myocardial infarction and/or stroke was associated with elevated plasma levels of homocysteine, and low plasma levels of folate, vitamins B12 and B6.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-09; Study Completion 1999-03